CLINICAL TRIAL: NCT07248358
Title: The Efface of Ketamine vs. Magnesium Sulphate in the Management of Pain After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: The Efface of Ketamine vs. Magnesium Sulphate in the Management of Pain After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Mustafa Hussain Imam, Mustafa Hussain Imam, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1096-2024-LNH-ERC
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Cholecystectomy Surgery; Postoperative Pain Management
Keywords: ketamine; magnesium sulphate; Laparoscopic Cholecystectomy; Pain; Postoperative Pain; Anesthesia
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Active Comparator): The ketamine dose was prepared at 0.5 mg/kg of body weight, diluted with normal saline to make a total volume of 10 mL, and administered intravenously as a single bolus during anesthesia reversal after the surgery was completed.
  Interventions: Drug: IV ketamine 0.5 mg/kg
- Magnesium Sulphate (Active Comparator): The magnesium sulfate dose was prepared as 2 mg, diluted with normal saline to a total volume of 10 mL, and administered intravenously as a single stat dose at the time of anesthesia reversal after completion of surgery.
  Interventions: Drug: IV 2mg of Magnesium Sulphate

INTERVENTIONS:
Drug: IV ketamine 0.5 mg/kg — Here is a rewritten and unbolded version of your paragraph:
  ---
  Patients in the ketamine group were given intravenous ketamine at a dose of 0.5 mg/kg of body weight, diluted with normal saline to a total volume of 10 mL. The solution was administered as a single intravenous injection at the time of anesthesia reversal, immediately after completion of laparoscopic cholecystectomy. The drug was given under aseptic conditions by an anesthetist who was unaware of group allocation. All patients received standard postoperative care, including intravenous diclofenac sodium 75 mg every 8 hours for baseline analgesia and intravenous ondansetron 4 mg for nausea prophylaxis. Postoperative pain was assessed at 1, 6, 12, and 24 hours using the Visual Analogue Scale (VAS). Patients reporting significant pain were given intravenous Kinz 5 mg as rescue analgesia, with the timing of administration recorded.
  Arms: Ketamine Group
Drug: IV 2mg of Magnesium Sulphate — Patients in the magnesium sulfate group received 2 mg of the drug, which was diluted with normal saline to a total volume of 10 mL and administered intravenously as a single stat dose at the time of anesthesia reversal following completion of laparoscopic cholecystectomy. The injection was performed under aseptic conditions by an anesthetist who was blinded to group assignment. All participants received routine postoperative care, including intravenous diclofenac sodium 75 mg every 8 hours for baseline pain control and intravenous ondansetron 4 mg to prevent nausea. Postoperative pain intensity was measured using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours. Patients experiencing significant pain were given intravenous Kinz 5 mg as rescue analgesia, and the timing of administration was recorded for documentation.
  Arms: Magnesium Sulphate

SUMMARY:
This prospective interventional study was conducted at Liaquat National Hospital and Medical College to compare the postoperative analgesic effects of ketamine and magnesium sulphate in patients undergoing laparoscopic cholecystectomy. A total of 78 ASA I-II patients were included and randomly allocated into two equal groups (39 patients in each group) using a sealed-envelope technique. One group received ketamine, while the other received magnesium sulphate, following a standardized intraoperative anesthesia protocol. All patients were provided routine postoperative medications according to institutional practice. Pain scores were recorded using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours after surgery. The objective of this study was to determine which drug offered better postoperative pain relief, thereby contributing to improved analgesic strategies for patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Effective postoperative pain control plays a crucial role in accelerating recovery, minimizing physiological stress, and improving patient satisfaction after laparoscopic cholecystectomy. This prospective interventional study was carried out in the Department of Anesthesiology at Liaquat National Hospital and Medical College to evaluate and compare the analgesic benefits of intravenous ketamine and magnesium sulphate in adults undergoing elective laparoscopic cholecystectomy.

A total of 78 patients classified as ASA I and II with uncomplicated symptomatic gallstones were recruited after obtaining ethical approval and written informed consent. The study was conducted in a double-blinded, participants were randomized into two groups through a sealed-envelope technique: Group K (n = 39) received ketamine, while Group M (n = 39) received magnesium sulphate adding both of the intervention were active drug agent. Patients with ASA III-V, chronic pain disorders, psychiatric illness, pregnancy or breastfeeding status, significant hepatic, renal, or cardiac impairment, or recent use of opioids or NSAIDs were excluded.

All enrolled individuals underwent routine preoperative evaluation and overnight fasting. General anesthesia was induced with propofol and atracurium and maintained with isoflurane, with continuous monitoring of vital parameters including heart rate, non-invasive blood pressure, ECG, oxygen saturation, and end-tidal CO₂. At the completion of surgery, neuromuscular blockade was reversed with neostigmine. Standard postoperative medications consisted of intravenous diclofenac sodium every 8 hours for background analgesia, along with ondansetron for nausea prophylaxis.

Postoperative pain levels were documented using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours following surgery. Patients who experienced significant pain were administered intravenous Kinz 5 mg as rescue analgesia, with administration times recorded by nursing personnel.

This study offered meaningful evidence regarding the comparative analgesic performance of ketamine and magnesium sulphate in the early postoperative period after laparoscopic cholecystectomy. The findings support their potential utility as part of a multimodal analgesic approach aimed at improving patient comfort and enhancing postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II. Elective laparoscopic cholecystectomy planned under general anesthesia. Normal baseline renal, hepatic, and coagulation profile. Able to give informed consent and communicate pain scores. Negative pregnancy test for women of childbearing age.

Exclusion Criteria:

* Allergy or hypersensitivity to ketamine, magnesium sulphate, or related drugs. History of psychiatric illness or substance abuse. Chronic use of opioids, benzodiazepines, or MAO inhibitors. Pregnant or breastfeeding women. Chronic pain disorders or use of analgesics within 7 days pre-op. Major hepatic, renal, or cardiovascular dysfunction. History of myopathy or seizure disorders. Patients with atrioventricular block or on calcium-channel blockers. Conversion to open cholecystectomy during surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | Postoperative pain was assessed at the 1st, 6th, 12th, and 24th hours
  Postoperative pain was evaluated using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours after surgery to compare the efficacy and duration of analgesia between the ketamine and lidocaine groups. These time points were chosen to capture both early and late pain responses within the first 24 hours of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asgher, Mbbs, FCPS, Study Director — Liaquat National Hospital
Locations (1):
- Anesthesiology Department Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No